CLINICAL TRIAL: NCT04015050
Title: A Randomised, Controlled, Double-blind, Parallel Group, Multi-country Study to Investigate the Safety and Tolerance of Infant Formula With Prebiotics and Postbiotics in Healthy Term Infants.
Brief Title: Randomised, Controlled Study to Assess Safety and Tolerance of Infant Formula With Prebiotics and Postbiotics in Healthy Infants.
Acronym: WAVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nutricia Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: EBB18FI23464
Record Dates: First submitted 2019-07-04; First posted 2019-07-10 (Actual); Last update posted 2021-12-17 (Actual); Status verified 2021-12

CONDITIONS: Healthy Term Infants

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test product (Experimental): Cow's milk based infant formula containing prebiotics and postbiotics
  Interventions: Other: milk based infant formula
- Control product (Active Comparator): Cow's milk based infant formula without prebiotics and postbiotics
  Interventions: Other: milk based infant formula

INTERVENTIONS:
Other: milk based infant formula — Cows milk ased infant formula

SUMMARY:
A randomised, controlled, double-blind, parallel group, multi-country study to investigate the safety and tolerance of infant formula with prebiotics and postbiotics in healthy term infants.

ELIGIBILITY:
Inclusion Criteria:

* 1. Healthy, singleton, term infants (gestational age ≥37 weeks + 0 days and ≤41weeks + 6 days);

  2. Infants with age at screening ≤14 days;

  3. Birth weight within 10th to 90th percentile per gestational age and sex, according to Intergrowth Standards;

  4. Head circumference at screening within ±2 SD per age and sex according to WHO Child Growth Standards;

  5. a Randomised groups: Infants who are exclusively formula fed and/or whose mothers have autonomously decided to exclusively formula feed, i.e. not to breastfeed or have ended breastfeeding before screening, and who are intending to exclusively formula feed at least till their infant is 17 weeks of age; OR b Breastfed reference group: Infants who are exclusively breastfed and whose mothers are intending to exclusively breastfeed at least till their infant is 17 weeks of age;

  6. Written informed consent from parent(s) and/or legal guardian(s) aged ≥18 years at screening.

Exclusion Criteria:

* 1. Randomised groups: Infants who require a special diet other than non-hydrolysed, cow's milk based infant formula (e.g. due to known or suspected to have cow's milk allergy, soy allergy and/or lactose intolerance);

  2. Infants with current or previous illnesses/conditions and/or known or suspected congenital diseases or malformations which could interfere with the study or its outcome parameters, such as but not limited to: GI malformations, congenital metabolic disorders, severe congenital cardiac disorders, immunodeficiency or major surgery, as per the clinical judgement of the Investigator;

  3. Infants with previous, current or intended participation in any other clinical study involving investigational or marketed products;

  4. Incapability of infants' parents to comply with study protocol as per the judgement of the Investigator;

  5. Infants born from mothers known to have (any) hepatitis or human immunodeficiency virus;

  6. Infants born from mothers with significant medical conditions during pregnancy that might interfere with the study or its outcome parameters or known to affect intra-uterine growth (e.g. placenta previa, pre-eclampsia, eclampsia, Type 1, 2 diabetes) as per clinical judgement of the Investigator;

  7. Infants born from mothers, who did participate in any clinical study involving investigational products during pregnancy, and for infants in Breastfed reference group: mothers who are currently participating or intend to participate in any clinical study involving investigational products during lactation.

Ages: 0 Days to 17 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 279 (Actual)
Dates: Start 2019-07-10 (Actual); Primary Completion 2021-12-03 (Actual); Study Completion 2021-12-03 (Actual)

PRIMARY OUTCOMES:
Weight gain | 17 weeks
  from baseline until the age of 17 weeks (test product versus control product). Weight gain will be calculated as weight (in grams) at visit minus weight at baseline divided by the number of days.

CONTACTS AND LOCATIONS:
Locations (1):
- Poliklinika Ginekologiczno-Położnicza Sp. z o.o. Sp. k., Bialystok, Poland

IPD SHARING:
Plan to Share IPD: Undecided